CLINICAL TRIAL: NCT03455751
Title: Precision Pain Management for Major Abdominal Surgery in Colorectal Surgery
Acronym: PPaM
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Failed to meet enrollment goals
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, David Liska, Associate Staff, Colorectal Surgery, The Cleveland Clinic
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 17-1540
Record Dates: First submitted 2018-02-28; First posted 2018-03-07 (Actual); Last update posted 2019-03-18 (Actual); Status verified 2019-03

CONDITIONS: Colorectal Cancer; Diverticular Disease; Crohn Disease; Ulcerative Colitis
Keywords: Pain Management; Pharmacogenomics
MeSH Terms: conditions — Colorectal Neoplasms; Diverticular Diseases; Crohn Disease; Colitis, Ulcerative; Agnosia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): The control arm will receive no intervention and will follow standard of care for post-operative pain management.
- PGx-guided (Experimental): The PGx-guided arm will received altered post-operative pain management based on the results of pharmacogenomic testing.
  Interventions: Genetic: PGx-guided post-operative pain management

INTERVENTIONS:
Genetic: PGx-guided post-operative pain management — Post-operative pain management as indicated by pharmacogenomic testing results.
  Arms: PGx-guided

SUMMARY:
The primary objectives of this study are to evaluate the potential for preoperative pharmacogenomics (PGx) testing to positively influence postoperative opioid use through visual analog scale (VAS) guided administration of narcotic equivalent and lower pain scores as measured by OBAS in patients undergoing major abdominal surgery.

ELIGIBILITY:
Inclusion Criteria:

* Subject capable of giving consent
* Age 18-80
* Scheduled for open colorectal resection at Cleveland Clinic main campus (with preoperative appointment scheduled at least five days before date of surgery)

Exclusion Criteria:

* Patient does not speak English
* Patient with substance-use disorder (including alcohol)
* Patient diagnosed with major depression
* Patient currently taking opioids
* Previous long-term opioid use (> 3 months)
* Previous opioid use with a dose of >100 milligram morphine equivalent (MME)
* Patient has pain-related disorder (e.g. fibromyalgia, sympathetic dystrophy, etc.)
* Documented allergy to pain medication

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2018-04-17 (Actual); Primary Completion 2019-01-09 (Actual); Study Completion 2019-01-09 (Actual)

PRIMARY OUTCOMES:
Post-operative opioid use | Post-op day 1
  Post-operative opioid use through visual analog scale guided administration of narcotic equivalent
Overall Benefit of Analgesia Score (OBAS) | Post-op day 1

SECONDARY OUTCOMES:
Length of stay | 30 days
Readmission rate | 30 days
Functional status | 4 weeks and 3 months
  Assessed through Duke Activity Status Index (DASI)

CONTACTS AND LOCATIONS:
Overall Officials: David Liska, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States